CLINICAL TRIAL: NCT02444689
Title: EMPower: Electronic Media Powering Positive Health Changes in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00065277; 1K23HL119622-01A1 (NIH)
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Hypertension; Prehypertension; Overweight; Obesity; Hypertrophy, Left Ventricular
Keywords: Blood pressure; Cardiovascular disease; Children; Adolescent; Pediatrics; End-organ damage
MeSH Terms: conditions — Hypertension; Prehypertension; Overweight; Obesity; Hypertrophy, Left Ventricular; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electronic Media Application (Experimental): Participants will receive an age-appropriate behavioral intervention designed to promote weight loss, improved diet quality, and exercise.
  Interventions: Behavioral: Electronic Media Application
- Control (Active Comparator): Participants will receive standard of care education and feedback on how to implement a heart healthy lifestyle to promote weight loss, improved diet quality and exercise.
  Interventions: Behavioral: Standard of care education

INTERVENTIONS:
Behavioral: Electronic Media Application — Children in the intervention group will receive motivation, education and coaching regarding therapeutic lifestyle changes via a smart phone electronic media application.
  Arms: Electronic Media Application
Behavioral: Standard of care education
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a technology-based behavioral Healthy Lifestyle intervention on adiposity (body mass index z-score), blood pressure (mean clinic systolic BP), and heart size (LVM) in comparison to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or Obese
* Speaks English

Exclusion Criteria:

* No smart phone / smart phone data plan
* Not willing to send/ receive text messages or download and use the study applications
* Neurological impairment/ developmental delay
* New / changes in anti-hypertensive medication or medication known to affect blood pressure within the last 6 months
* Prior diagnosis of congenital heart disease or cancer
* Pregnancy
* Taking medication with weight gain as a side effect
* Taking medications for weight loss/ participation in another weight loss program

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2015-07; Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Change in adiposity as measured by change in BMI z-score | 6 months from date of randomization

SECONDARY OUTCOMES:
Change in clinic systolic blood pressure | 6 months from date of randomization
Change in left ventricular mass index | 6 months from date of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Tammy M Brady, M.D., Ph.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States